CLINICAL TRIAL: NCT04711486
Title: A Single-centre, Randomized, Placebo-controlled, Double-blind, Phase 1b Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Contraloid Acetate in Patients With Mild Cognitive Impairment Due to Alzheimer's Disease
Brief Title: Evaluation of Safety of Contraloid Acetate in Patients With Mild Cognitive Impairment Due to Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Berlin Institute of Health (Other); Federal Agency for Disruptive Innovation - SPRIN-D (Unknown)
Responsible Party: Principal Investigator, Oliver Peters, MD, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ContraloidAD
Record Dates: First submitted 2020-12-15; First posted 2021-01-15 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Mild Cognitive Impairment Due to Alzheimer's Disease
MeSH Terms: interventions — microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contraloid acetate (Experimental): 300 mg Contraloid/participant administered orally (for 28 days) as a single daily dose.
  Other Name: PRI-002
  Interventions: Drug: Contraloid acetate
- Placebo (Placebo Comparator): 300 mg Placebo (Microcrystalline cellulose)/participant administered orally (for 28 days) as a single daily dose.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Contraloid acetate — Oral administration of drug substance capsules
  Other Names: PRI-002
  Arms: Contraloid acetate
Drug: Placebo — Oral administration of placebo without any exipients.
  Other Names: Microcrystalline cellulose
  Arms: Placebo

SUMMARY:
Patients with mild cognitive impairment due to Alzheimer's disease (MCI due to AD) are at high risk to develop Alzheimer´s dementia. The therapeutic agent Contraloid has the potential to influence the chronic neurodegenerative process of AD. As Contraloid was so far only administered to healthy subjects, the rational of the proposed study is first to collect safety data in patients diagnosed with MCI due to AD, as the absorption, distribution, metabolism and excretion processes may be altered by disease, aging, comorbidities and concomitant drug therapies. Additionally, the design of a subsequent phase II study will be based on the data of this study. The results of the exploratory analyses will enable power calculations and the identification of the most useful and reliable biomarkers for the subsequent proof of concept phase II study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with MCI due to AD according to DSM-V
2. Age between 50 and 80 years (male and female)
3. MMSE score 22-30
4. Written informed consent (according AMG §40 (1) 3b)
5. Level of Aβ-oligomers: mind. 1fM
6. CSF according to diagnosis (p-tau > 62 pg/ml, total CSF Aβ 1-42/1-40 ratio ≤ 0.055)
7. 3 months prior to screening stable medication
8. Females without childbearing potential

Exclusion Criteria:

1. History of seizures
2. History of stroke or TIA
3. Unstable medical, neurological or psychiatric condition
4. Current treatment with one of the following substances:

   * Typical antipsychotic or neuroleptic medication within 6 months of screening
   * Anti-coagulation medications within 3 months of screening
   * Chronic use of opiates or opioids (including long-acting opioid medication) within 3 months of screening
   * Stimulant medications (amphetamine, methylphenidate preparations, or modafinil) within 1 month of screening and throughout the study
   * Chronic use of benzodiazepines, barbiturates, or hypnotics from 3 months before screening
5. Persons who are legally detained in an official institution
6. Persons who may be dependent on the sponsor, the investigator or the trial site
7. Persons without caregiver
8. Participation in other clinical trials according to AMG (1 month before the time of this trial)
9. Persons showing EEG abnormalities

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2022-01-13 (Actual); Study Completion 2022-01-13 (Actual)

PRIMARY OUTCOMES:
Safety: Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | From baseline (day 1) to follow-up (day 56)
  Number of Adverse Events
Safety: Number of Participants with abnormal laboratory values (urinalysis, CBC, Quick, PTT, Creatinine, CK, CRP, ALT, AST) | From baseline (day 1) to follow-up (day 56)
  Laboratory values: urinalysis, CBC, Quick, PTT, Creatinine, CK, CRP, ALT, AST
Safety: Number of Participants with abnormal ECG values | From baseline (day 1) to follow-up (day 56)
  ECG

SECONDARY OUTCOMES:
Pharmacokinetics: Peak Plasma Concentration (Cmax) | pre-dose and 15 min, 1 hour, 2 hours, 4 hours post-dose at day 1 and day 28
  Cmax in plasma
Pharmacokinetics: The time at which Cmax is observed (Tmax) | pre-dose and 15 min, 1 hour, 2 hours, 4 hours post-dose at day 1 and day 28
  Tmax in plasma
Pharmacokinetics: Terminal elimination half-life (t1/2) in plasma | pre-dose and 15 min, 1 hour, 2 hours, 4 hours post-dose at day 1 and day 28
  t1/2 in plasma

OTHER OUTCOMES:
Efficacy: Change of biomarkers in CSF | Baseline to end of treatment (day 28) to follow-up (day 56)
  Biomarkers: p-tau, t-tau, NFL, Aβ 1-40, Aβ 1-42 and Aβ and tau oligomers
Efficacy: Change of biomarkers in plasma | Baseline to end of treatment (day 28) to follow-up (day 56)
  Biomarkers: p-tau, t-tau, NFL, Aβ 1-40, Aβ 1-42 and Aβ and tau oligomers
Efficacy optional: Change of biomarkers in feces | Baseline to end of treatment (day 28) to follow-up (day 56)
  Biomarkers: p-tau, t-tau, NFL, Aβ 1-40, Aβ 1-42 and Aβ and tau oligomers
Efficacy: Change in CERAD+ test battery scores | Baseline to end of treatment (day 28) to follow-up (day 56)
Efficacy: Change in CDR-Sum of boxes | Baseline to end of treatment (day 28) to follow-up (day 56)

CONTACTS AND LOCATIONS:
Locations (1):
- Charité University Medicine, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kutzsche J, Cosma NC, Kauselmann G, Fenski F, Bieniek C, Bujnicki T, Pils M, Bannach O, Willbold D, Peters O. Oral PRI-002 treatment in patients with MCI or mild AD: a randomized, double-blind phase 1b trial. Nat Commun. 2025 May 6;16(1):4180. doi: 10.1038/s41467-025-59295-z. PMID 40324978